CLINICAL TRIAL: NCT05184530
Title: In-hospital Initiation of PCSK9 Inhibitor and Short-term Lipid Profile Alteration, as Well as In-hospital Mortality and Readmission Rate in Patients With Acute Myocardial Infarction
Brief Title: In-hospital Initiation of PCSK9 Inhibitor in Patients With Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, She JianQing, First Affiliated Hospital Xi'an Jiaotong University, First Affiliated Hospital Xi'an Jiaotong University
Other Study IDs: 82100477-1
Record Dates: First submitted 2022-01-05; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease | interventions — evolocumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Statin Group: AMI patients with Statin therapy.
- Ezetimibe Group: AMI patients with Statin plus Ezetimibe therapy.
- PCSK9i Group: AMI patients with Statin plus PCSK9i therapy.
  Interventions: Drug: Evolocumab 140 MG/ML
- Triple Group: AMI patients with Statin plus Ezetimibe plus PCSK9i therapy
  Interventions: Drug: Evolocumab 140 MG/ML

INTERVENTIONS:
Drug: Evolocumab 140 MG/ML — 140 mg per two weeks, subcutaneous injection
  Groups: PCSK9i Group; Triple Group

SUMMARY:
Proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitors have been shown to improve cardiovascular outcomes when added to conventional statin therapy. This study aims to investigate the efficacy and safety of in-hospital initiation of PCSK9 inhibitor among patients with acute myocardial infarction(AMI) based on real-world experience.

A total of 7556 AMI patients from the biobank database between January 2016 and December 2020 were screened for eligibility. After excluding those without revascularization or Statin based therapy, the remaining 5802 Statin users, 801 Statin plus Ezetimibe users and 170 Statin plus Evolocumab users (including 95 users without and 75 users with Ezetimibe), were selected for this study. Then, 1st and 3rd-month follow-up data were collected and analysed, including in-hospital mortality, readmission rate and lipid profiles

ELIGIBILITY:
Inclusion Criteria:

* confirmed admission diagnosis of AMI and were defined based on the universal definition criteria by the American Cardiology College

Exclusion Criteria:

* (1) severe noncardiac disease with an expected survival of less than 1 year and unwillingness to participate; (2) patients over the age of 80 years or living far away from the hospital's catchment area.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 7556 consecutive patients admitted to the cardiology department of the First Affiliated Hospital of Xi'an Jiaotong University for AMI between January 2016 and December 2020 were enrolled.
Sampling Method: Probability Sample
Enrollment: 7556 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Readmission rate | 1 YEAR

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lou B, Liu H, Luo Y, Jiang GT, Wu H, Wang C, Wu Y, Zhou B, Yuan Z, She J, Liu J. In-hospital initiation of PCSK9 inhibitor and short-term lipid control in patients with acute myocardial infarction. Lipids Health Dis. 2022 Oct 24;21(1):105. doi: 10.1186/s12944-022-01724-9. PMID 36280861